CLINICAL TRIAL: NCT05427643
Title: Evaluation of Secondary Dental Implant Stability Utilized For Narrow Ridges With Injectable Platelet Rich Fibrin Versus Straightforward Cases
Brief Title: Evaluation of the Effect of Injectable Platelet Rich Fibrin on Stability of Dental Implant for Narrow Ridges
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sora Salam Majeed (Other)
Responsible Party: Sponsor-Investigator, Sora Salam Majeed, Principle investigator, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 964_07706223546
Record Dates: First submitted 2022-06-17; First posted 2022-06-22 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Dental Implantation, Endosseous
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): patients need dental implants with narrow alveolar ridge of less than 6 mm horizontal width .
  they will receive dental implants with I_PRF mixed with synthetic bone graft.
  Interventions: Procedure: study group
- control group (Experimental): patients need dental implant with adequate horizontal bone with of more than 6 mm.
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: study group — dental implant procedure under local anesthesia
  Other Names: I-PRF preparation
  Arms: study group
Procedure: control group — dental implant procedure under local anesthesia
  Arms: control group

SUMMARY:
the main aim of the study is to evaluate the secondary implant stability when using dental implants with injectable platelet rich fibrin accompanied by non-autogenous bone graft material in narrow ridge cases versus straightforward ridges , in clinical comparative study.

DETAILED DESCRIPTION:
the main aim of the study is to evaluate the secondary implant stability when using dental implants with injectable platelet rich fibrin accompanied by non-autogenous bone graft material in narrow ridge cases versus straightforward ridges , in clinical comparative study.

Study design:

Forty implants will be installed for this prospective clinical study, the implants will be equally divided into two groups.

Group A (control group) in which the implants will be installed in a straightforward cases.

Group B (study group) in which the implants will be installed by utilizing injectable PRF with non-autogenous bone graft material in narrow ridges.

Preparation of Injectable Platelet Rich Fibrin for the narrow ridge cases is as following:

Five ML of autologous blood to be collected from the forearm (median cubital vein \ cephalic vein \ basilic vein ) by needle gauge with a 5mL sterile syringe without anticoagulant. The entire blood is moved to a 5 milliliter plastic tube, directly centrifugated for 3 minutes at 700 rpm/min at room temperature. A liquid form ( Injectable PRF ) is then achieved on top of the tube just and the red corpuscles at the bottom. Subsequently, the Injectable PRF liquid form is collected from the tube by a sterile plastic syringe, Then it will be mixed with non-autogenous bone graft waiting for 4min, and applied in the area with narrow ridge( deficiency in the horizontal bone width ) .

Follow up Twenty four weeks after surgery , The uncoverage surgery is done under L.A using a tissue paunch for installing the healing abutment ( gingival former ) , Then the secondary stability of implant (Osseointegration) is to be measured using the (Anycheck ) device , and comparing the 2 groups

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age.
2. Absence of general medical contraindications for oral surgery procedures such as (Radiated jaws / uncontrolled Diabetic patient / uncontrolled hypertensive patient ).
3. Straightforward cases / narrow ridges (less than 6mm horizontal bone width) according to SAC classification ( advanced surgery ) cases.
4. Patients with reasonable oral hygiene.
5. Partially or totally edentulous alveolar ridges.

   -

Exclusion Criteria:

1. Uncontrolled medically compromised patients such as : (heart diseases uncontrolled blood pressure, endocrine disorders such as (diabetes , Thyroid disorders , osteoporosis ) , immuno-compromised patient and any condition influence bone healing ……etc.
2. Heavy smokers ( ≥ 20 cigarettes a day).
3. Patients with parafunctional habits.
4. Complicated cases according to SAC classification.
5. Patient with signs of acute infection and purulent exudates at the site of implant placement as revealed by clinical and radiographical examination.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
secondary implant stability | six months
  measured by Anycheck device after osseointegration time

CONTACTS AND LOCATIONS:
Locations (1):
- college of dentistry university of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The application of injectable platelet-rich fibrin in regenerative dentistry: A systematic scoping review of In vitro and In vivo studies — http://pubmed.ncbi.nlm.nih.gov/35368368/